CLINICAL TRIAL: NCT04654169
Title: Effectiveness of Suprascapular Nerve Block in Addition to Intra-articular Corticosteroid Injection in Adhesive Capsulitis: A Double-blind, Randomized Controlled Trial
Brief Title: Suprascapular Nerve Block in Addition to Intra-articular Corticosteroid Injection in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Kardelen Gencer Atalay, Principal Investigator, Marmara University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2018.836
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Adhesive Capsulitis of the Shoulder
Keywords: Adhesive Capsulitis of the Shoulder; Intra-Articular Injections; Nerve Blockade
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized controlled trial, to have two groups with a single arm
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation information of patients was only given to the physiatrists who would apply the intervention. Another physiatrist who completed the pre and post-treatment assessments and the patients were blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The IAI and SSNB group (Experimental): Ultrasound-guided IAI and SSNB are planned to apply by at least three-year experienced physiatrists. Patients are planned to initiate a six-week rehabilitation program supervised by the same physiotherapist one day after the intervention.
  Interventions: Procedure: Ultrasound-guided IAI; Procedure: Ultrasound-guided SSNB
- The only-IAI group (Active Comparator): Ultrasound-guided IAI is planned to apply by at least three-year experienced physiatrists. Patients are planned to initiate a six-week rehabilitation program supervised by the same physiotherapist one day after the intervention.
  Interventions: Procedure: Ultrasound-guided IAI

INTERVENTIONS:
Procedure: Ultrasound-guided IAI — Ultrasound-guided IAI was applied with a posterior glenohumeral joint in-plane injection technique.
Procedure: Ultrasound-guided SSNB — Ultrasound-guided SSNB was carried out with a supraspinatus fossa level in-plane injection technique
  Arms: The IAI and SSNB group

SUMMARY:
Adhesive capsulitis is a disease that negatively affects a person's quality of life by causing severe pain and limitation in the movements of the shoulder joint in all directions. Conservative approaches including nonsteroidal anti-inflammatory drugs or oral corticosteroid usage and physiotherapy program are the first choice for the treatment. However, painful exercises usually prevent patients from fully participating in the physiotherapy program. For this reason, interventional procedures such as intra-articular corticosteroid injection (IAI) and suprascapular nerve block (SSNB) are preferred to be applied before the physiotherapy program.

The aim of this study is to reveal both short and long-term effects of SSNB and IAI combination on pain, shoulder range of motion (ROM), disability, and quality of life in patients with adhesive capsulitis. It is hypothesized that the addition of SSNB to IAI results in greater improvements in pain, passive and active shoulder ROMs, disability, and quality of life.

DETAILED DESCRIPTION:
Adhesive capsulitis (AK), also known as frozen shoulder, is a disease that negatively affects a person's quality of life by causing severe pain and limitation in the movements of the shoulder joint in all directions. Although the underlying etiology is not clear, it may develop as a result of primary (idiopathic) or secondary causes such as diabetes mellitus, malignancy, thyroid dysfunction, hypoadrenalism, Parkinson's disease, stroke, cardiac and pulmonary diseases, or local shoulder problems such as trauma, tendinitis, rupture. Prolonged immobilization after injuries is another important risk factor for adhesive capsulitis. It is more common in women between the ages of 40-60. Conservative approaches including nonsteroidal anti-inflammatory drugs or oral corticosteroid usage and physiotherapy program are the first choice for the treatment. The physiotherapy program consisting range of motion (ROM), stretching and strengthening exercises are often painful and prevent the patient's full participation. For this reason, interventional procedures such as intra-articular corticosteroid injection (IAI) and suprascapular nerve block (SSNB) are preferred to be applied before the physiotherapy program.

The aim of this study is to reveal both short and long-term effects of SSNB and IAI combination on pain, shoulder ROM, disability, and quality of life in patients with adhesive capsulitis. It is hypothesized that the addition of SSNB to IAI results in greater improvements in pain, passive and active shoulder ROMs, disability, and quality of life. The primary outcome measure of the study is determined to be the Shoulder Pain and Disability Index (SPADI), while the secondary outcome measures to be the Numeric Rating Scale (NRS), active and passive ROMs, and the Short Form 36 (SF-36).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of adhesive capsulitis
* Bening of symptoms at least three months prior
* Having shoulder pain with passive ROM limitation greater than 30° compared to normal values in at least two directions

Exclusion criteria were:

* Adhesive capsulitis stages 3 and 4
* Previous trauma, IAI, or surgery history
* Evidence of complete rotator cuff tear, calcific tendinitis, biceps tendinitis, glenohumeral or acromioclavicular arthritis on magnetic resonance imaging
* Uncontrolled diabetes mellitus
* Known coagulation disorder
* Contraindication to corticosteroid or local anesthetic injection.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Baseline (T0)
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire consisting of 13 items divided into two subscales varying between 0 to 100, with a higher value indicating worse condition.
Shoulder Pain and Disability Index (SPADI) | Three weeks after the intervention (T2)
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire consisting of 13 items divided into two subscales varying between 0 to 100, with a higher value indicating worse condition.
Shoulder Pain and Disability Index (SPADI) | Three months after the intervention (T3)
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire consisting of 13 items divided into two subscales varying between 0 to 100, with a higher value indicating worse condition.
Shoulder Pain and Disability Index (SPADI) | Twelve months after the intervention (T4)
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire consisting of 13 items divided into two subscales varying between 0 to 100, with a higher value indicating worse condition.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | Baseline (T0)
  Numeric Rating Scale (NRS) is used to grade pain intensity between 0 (no pain) to 10 (worst pain) by the patient.
Numeric Rating Scale (NRS) | One hour after the intervention (T1)
  Numeric Rating Scale (NRS) is used to grade pain intensity between 0 (no pain) to 10 (worst pain) by the patient.
Numeric Rating Scale (NRS) | Three weeks after the intervention (T2)
  Numeric Rating Scale (NRS) is used to grade pain intensity between 0 (no pain) to 10 (worst pain) by the patient.
Numeric Rating Scale (NRS) | Three months after the intervention (T3)
  Numeric Rating Scale (NRS) is used to grade pain intensity between 0 (no pain) to 10 (worst pain) by the patient.
Numeric Rating Scale (NRS) | Twelve months after the intervention (T4)
  Numeric Rating Scale (NRS) is used to grade pain intensity between 0 (no pain) to 10 (worst pain) by the patient.
Short Form-36 | Baseline (T0)
  Short Form-36 (SF-36) is a widely-used and well-documented health-related quality of life index. The SF-36 consists of 36 questions; It survey has eight sub-dimensions, including physical functioning, role limitations due to physical problems, pain, general health perception, mental health, role limitations due to emotional problems, vitality, and social functioning, which are evaluated individually. A higher score on a 0-100 scale indicates a better quality of life.
Short Form-36 | Three weeks after the intervention (T2)
  Short Form-36 (SF-36) is a widely-used and well-documented health-related quality of life index. The SF-36 consists of 36 questions; It survey has eight sub-dimensions, including physical functioning, role limitations due to physical problems, pain, general health perception, mental health, role limitations due to emotional problems, vitality, and social functioning, which are evaluated individually. A higher score on a 0-100 scale indicates a better quality of life.
Short Form-36 | Three months after the intervention (T3)
  Short Form-36 (SF-36) is a widely-used and well-documented health-related quality of life index. The SF-36 consists of 36 questions; It survey has eight sub-dimensions, including physical functioning, role limitations due to physical problems, pain, general health perception, mental health, role limitations due to emotional problems, vitality, and social functioning, which are evaluated individually. A higher score on a 0-100 scale indicates a better quality of life.
Short Form-36 | Twelve months after the intervention (T4)
  Short Form-36 (SF-36) is a widely-used and well-documented health-related quality of life index. The SF-36 consists of 36 questions; It survey has eight sub-dimensions, including physical functioning, role limitations due to physical problems, pain, general health perception, mental health, role limitations due to emotional problems, vitality, and social functioning, which are evaluated individually. A higher score on a 0-100 scale indicates a better quality of life.
Shoulder range of motion (ROM) evaluated with a handheld goniometer | Baseline (T0)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, internal and external rotation.
Shoulder range of motion (ROM) evaluated with a handheld goniometer | One hour after the intervention (T1)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, internal and external rotation.
Shoulder range of motion (ROM) evaluated with a handheld goniometer | Three weeks after the intervention (T2)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, internal and external rotation.
Shoulder range of motion (ROM) evaluated with a handheld goniometer | Three months after the intervention (T3)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, internal and external rotation.
Shoulder range of motion (ROM) evaluated with a handheld goniometer | Twelve months after the intervention (T4)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, internal and external rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Yagci, Prof, Study Director — Marmara University
Locations (1):
- Kardelen Gencer Atalay, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No